CLINICAL TRIAL: NCT06912685
Title: Pilot Test of an Innovative Implementation Strategy to Improve Reach, Quality, and Equity in Child Maltreatment Prevention
Brief Title: Pilot Test of Innovative Child Maltreatment (CM) Prevention Strategy
Acronym: (CM)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Hannah Espeleta, Research Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00141218
Record Dates: First submitted 2024-11-13; First posted 2025-04-06 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-04

CONDITIONS: Parenting Intervention; Maltreatment; Prevention
Keywords: Disease Prevention; Healthy Volunteer Studies; Infant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SafeCare as Usual (Active Comparator): Normal care is SafeCare, an evidence-based home visiting parenting program with three modules focused on child health, home safety, and parent-child relationships. SafeCare sessions typically occur weekly over 18 weeks.
  Interventions: Other: SafeCare
- Technology Enhanced Implementation Package (TEIP) (Experimental): The TEIP group will also receive SafeCare and the SafeCare provider will use added guidance on when to use in person or virtual sessions. They will also get access to different support tools, like games or videos, that may be played during online sessions.
  Interventions: Other: Technology Enhanced Implementation Package; Other: SafeCare

INTERVENTIONS:
Other: Technology Enhanced Implementation Package — The Technology Enhanced Implementation Package for SafeCare delivery consists of protocol adaptations, evidence-informed guidelines, and digital health resources to improve SafeCare outcomes related to reach, quality, and equity.
  Arms: Technology Enhanced Implementation Package (TEIP)
Other: SafeCare — SafeCare is an evidence-based home visiting parenting program with three modules focused on child health, home safety, and parent-child relationships. SafeCare sessions typically occur weekly over 18 weeks.

SUMMARY:
Millions of children are victims of maltreatment each year in the United States. Research on home visiting programs show that child maltreatment can be prevented; however, these programs struggle to reach families in need and provide high quality care. SafeCare is a sustainable and effective home visiting child maltreatment prevention program, serving over 8,000 families each year. This study will examine the feasibility and implementation of a hybrid in-person/virtual delivery model for SafeCare with 12 home visiting providers and 40 caregivers to inform how home visiting programs are delivered to maximize reach to families, improve family outcomes, and decrease harm to children.

DETAILED DESCRIPTION:
Child maltreatment (CM) is a public health priority, affecting millions of children each year. Evidence-based home visiting (HV) models are gold standard CM prevention programs that intervene on modifiable risk factors. Despite their effectiveness and national implementation, HV is resource intensive which limits their potential reach and impact. HV programs serve only 3% of high-risk families, with limited access for minoritized and rural-dwelling families. Rigorous research is needed to guide approaches to implementing HV to ensure agencies can deliver the highest-quality care with more accessibility and equity without compromising child safety. Preliminary data during the COVID-19 pandemic offered insight to the benefits of virtual, telehealth-based visits for CM prevention and enabled service agencies to observe that quality and safety concerns can be managed in most cases. The consensus of experts and HV providers is that hybrid, telehealth leveraged HV implementation can enhance access, quality, and efficiency of CM prevention models. Moreover, technology-based supports are needed to engage families, drive skill acquisition, support model fidelity, and improve accuracy in safety and skill assessment. Through an institutional KL2 award (PI: Espeleta), leveraging community advisory boards, secondary data analysis of clinical services data, and user-centered design methods, I am developing a telehealth-compatible, technology-enhanced, hybrid in-person/virtual implementation package for CM prevention. This package will consist of protocol adaptations, evidence-informed guidelines, and digital health resources to improve implementation outcomes related to reach, quality, and equity. However, the KL2 does not include a pilot RCT, which is essential to establish the feasibility of the implementation package as well as the RCT methodology in preparation for a future R01. The project's goals are to 1) Refine and preliminarily evaluate the TEIP and the feasibility of the research methodology with 12 providers and 40 families; and 2) Assess implementation factors related to the TEIP including its usability, acceptability, and feasibility with key constituents. Findings will inform a future R01 submission to evaluate the hybrid HV/virtual implementation on dimensions of equitable reach, effectiveness, implementation, and maintenance.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* English language proficiency
* Ability to provide informed consent for themselves
* Has at least one child between the ages of 0-5 years old - Caregivers Only
* Has completed at least 1 module of SafeCare since April 2021 - Caregivers Only
* SafeCare enrollment has been completed (e.g., not currently enrolled in SafeCare). - Caregivers Only
* Current employment at a SafeCare agency - Agency Leaders Only
* Full- or part-time employment at a SafeCare agency - Providers Only
* Must be fully certified to provide SafeCare services - Providers Only
* Must be providing services for at least 6 months - Providers Only

Exclusion Criteria:

* Evidence of significant cognitive disability, developmental delay, or pervasive developmental disorder that would prohibit capacity to consent for themselves - Caregivers Only
* There are no primary exclusion criteria for the Providers.
* There are no primary exclusion criteria for Agency Leaders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
SafeCare Sick or Injured Child Checklist | From the enrollment to the end the Health module, ~6 weeks after starting Health module
  As part of routine SafeCare delivery, providers assess caregiver scores on structured assessments that are part of the Child Health module. Assessments are conducted at the first and last session of this module and scores are recorded in the NSTRC Provider portal. Parents are presented with various health scenarios and respond with actions they would take during those scenarios. Scores represent the percentage of steps reported correctly across all scenarios.
Child Planned Activities Training Checklist | From the enrollment to the end the Parent Child Interaction module, ~6 weeks after starting Parent Child module
  As part of routine SafeCare delivery, providers assess caregiver scores on structured assessments that are part of the Parent-Child and Parent-Infant Interaction modules. Assessments are conducted at the first and last session of this module and scores are recorded scores in the NSTRC Provider portal. Providers rate parents on the number of interaction skills used during three different interactions with their child, with total scores representing the average percentage of skills used across the three interactions.
SafeCare Home Observation Checklist | From the enrollment to the end the Safety module, ~6 weeks after starting Safety module
  As part of routine SafeCare delivery, providers assess caregiver scores on structured assessments that are part of the Home Safety module. Assessments are conducted at the first and last session of this module and scores are recorded in the NSTRC Provider portal. Providers assess three commonly used rooms in the home and count the number of accessible safety hazards across all rooms.
Brief Child Abuse Potential Inventory | Baseline, 3- and 6-month follow up
  The BCAP is a 33-item caregiver self-report measure that assesses factors related to child abuse potential and underlying factors related to child abuse risk. The BCAP can be completed in less than 5 minutes, is made up of minimally intrusive items, and is written below a fourth grade reading level. It is a valid and reliable tool for assessing parenting risk.
Children Services Involvement | Baseline, 3- and 6-month follow up
  Caregivers will self-report on their interactions with child services during the study period. They will answer questions regarding the number of child welfare referrals received, any child placement changes, and current case status.

SECONDARY OUTCOMES:
Parent-Child Conflict Tactics Scale | Baseline, 3-month and 6-month follow up
  The CTS-PC is a 22-item caregiver self-report measure of parenting including neglect, physiological and physical maltreatment of children, and positive disciplinary strategies (e.g., non-violent discipline). Respondents are asked to reflect on their parenting behavior in the past year and rate items on a 7-point scale, with higher scores indicating greater frequency the parenting behavior.
Parenting Stress Inventory | Baseline, 3-month and 6-month follow up
  The PSI is a 36-item caregiver self-report scale designed to measure stressors in parenthood. There are three subscales with 12 items each including the dysfunctional interactions subscale, the difficult child subscale, and the parental distress subscale. Caregivers respond on a five-point scale with higher numbers indicating greater parenting stress.
Brief Symptom Inventory | Baseline, 3-month and 6-month follow up
  The BSI is a 53-item self-report symptom scale where caregivers will rate how much discomfort the problem presented in the item has caused them in the past seven days on a scale from 0 to 4. The measure includes subscales measuring nine symptoms. The Global Severity Index, a mean of all subscales, was used in this study. Test-retest reliability and internal consistency are very good.
Patient Health Questionnaire | Baseline, 3-month and 6-month follow up
  The PHQ-8 is widely used, 8-item screening tool for depression where caregivers will rate 8 symptoms on a four-point descriptive scale from 0 to 3. Criteria validity and internal validity have been established.
NIDA Quick Screen | Baseline, 3-month and 6-month follow up
  The NIDA Quick screen consists of four questions regarding the frequency of which respondents have used illegal drugs, prescription drugs for non-medical reasons, tobacco, or multiple drinks containing alcohol.
Social Provisions Scale | Baseline, 3-month and 6-month follow up
  The SPS is a 12-item self-report scale designed to measure overall perceived social support for adults.
Protective Factors Survey | Baseline, 3-month and 6-month follow up
  The PFS assesses five protective factors for child maltreatment including parenting knowledge, nurturing behaviors, and family functioning. Each domain includes four or five items and caregivers respond on a seven-point scale.
Family Resource Scale | Baseline, 3-month and 6-month follow up
  The FRS-revised is a 30-item self-report measure of the adequacy of resources in households with children. Items load on seven scales corresponding to income, childcare, communication/employment, intrafamily support, physical shelter, nutrition/protection, health/necessities, and growth/social support.
The Accountable Health Communities (AHC) Health-Related Social Needs (HRSN) Screening Tool | Baseline, 3-month and 6-month follow up
  The AHC HRSN screening tool is a 10-item self-report tool to help identify respondent needs on 5 core domains of housing instability, food insecurity, transportation problems, utility help needs, and interpersonal safety.
Client Satisfaction Survey | 3-month follow up
  The Client Satisfaction Survey is a short rating scale that assesses caregiver satisfaction with SafeCare content, the usefulness of training strategies and target skills, technology used during training, and a general rating of the home visitor. Items are rated on a. 5-point scale. Surveys are submitted by caregivers online following each SafeCare module completed.
Client Cultural Competency Inventory | 3-month follow up
  The CCCI is a caregiver self-report instrument reflecting their perception of the cultural competency of services. The instrument has a low susceptibility to social desirability bias and good internal consistency and temporal stability and has been used in mental health services utilization research.
Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure | 3-month follow up
  The AIM, IAM, and FIM measure is a self-report measure consisting of 15 items (5 items pers scale) that range from "completely disagree" to "completely agree." This measure can be tailored to your specific intervention to gather feedback on its acceptability, appropriateness, and feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Espeleta, Principal Investigator — Medical University of South Carolina

IPD SHARING:
Plan to Share IPD: No